CLINICAL TRIAL: NCT03263598
Title: Clinical Significance and Correlation Between the 24-Hour Urine Sodium Excretion and the Spot Urine Na/K Ratio in Cirrhotic Patients With Ascites.
Brief Title: Validation of Diagnostic Usefulness of the Random Urine Na/K Ratio for Replacement of 24hr Urine Na Excretion in Cirrhotic Patients With Ascites
Acronym: urine Na/K
Status: Completed | Type: Observational
Sponsor: Jang Byoung Kuk (Other)
Collaborators: Yeungnam University College of Medicine (Other); Kyungpook National University Hospital (Other); Daegu Catholic University Medical Center (Other); DongGuk University (Other)
Responsible Party: Sponsor-Investigator, Jang Byoung Kuk, Keimyung University Dongsan medical center, Keimyung University Dongsan Medical Center
Organization: Keimyung University Dongsan Medical Center (Other)
Other Study IDs: random Urine Na/K
Record Dates: First submitted 2016-08-18; First posted 2017-08-28 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Liver Cirrhosis; Ascites
Keywords: liver cirrhosis; ascites
MeSH Terms: conditions — Liver Cirrhosis; Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The low sodium intake is important for ascites control in liver cirrhosis patients. Therefore, World Health Organization (WHO) recommends reduction of sodium (Na) to 2g/day for adults. The 24-hour urine Na excretion has been regarded as a standard method to estimate the amount of daily dietary sodium intake. However, it is too inconvenient to apply to patients or the general population in practice. For this reason, it has been suggested that a spot urine Na/potassium (K) ratio could be replaced with the 24-hour urine Na excretion. However, the evidence is not sufficient for that. The investigators will evaluate the usefulness of spot urine Na/K ratio to estimate the dietary sodium intake. The investigators will also verify several formulas of estimating the 24-hour Na excretion with spot urine Na, K, Creatinine (Cr).

DETAILED DESCRIPTION:
● Detailed Description:

1. Measurements: they should be performed for 2 days (the urine collected within 24 hrs)

   * 24-hour urine Na, K and Creatinine (patients were instructed to collect all subsequent urine voids over the next 24-hour period including the ﬁrst void of the following day.)
   * Spot urine Na, K, Creatinine with the same urine sample in some containers provided to patients. (every urination)
2. Calculation

   * Na/K Ratio with spot urine Na, K
   * Estimating 24-hour urine Na with spot urine Na, K, Cr by using some formulas.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhotic patients with ascites diagnosed by imaging study, biopsy or clinically, regardless of taking diuretics.

Exclusion Criteria:

* Uncontrolled sepsis or systemic infection.
* Serum Creatinine >1.5 mg/dL.
* Patients who are being treated for cancers except hepatocellular carcinoma.
* Patients who refuse the examine or are not cooperative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers from the patient population including liver cirrhosis with ascites in multi-center.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2016-05; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the usefulness of urine Na / K ratio as a clinical indicator to replace the 24-hour urine sodium excretion (mEq/L) in liver cirrhosis patients with ascites. | After 24 hours of urine collection
  Previous studies have reported that the spot urine Na / K ratio is 90 percent accuracy compared to 24hr urine Na excretion. To verify this, measure spot urine Na, K (mEq/L) by using the same sample as the 24-hour sodium and creatinine excretion and confirm with receiver operator characteristic (ROC) curve to find the best cutoff point of spot urine Na / K ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Jang Byoung Kuk, Daegu, Kyoungpuk, South Korea

IPD SHARING:
Plan to Share IPD: Undecided